CLINICAL TRIAL: NCT01015599
Title: Healthy Opportunities for Physical Activity and Nutrition (HOP'N) After-School Project
Acronym: HOP'N
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kansas State University (Other)
Collaborators: Iowa State University (Other)
Responsible Party: David Dzewaltowski, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USDA no. 2005-35215-15418
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2009-11

CONDITIONS: Obesity Prevention
Keywords: Obesity prevention; after-school; physical activity; fruit; vegetable; children
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HOP'N After-School Program (Experimental): After-school program with daily physical activity following CATCH guidelines, daily fruit/vegetable snack, and weekly nutrition and physical activity education based on social cognitive theory.
  Interventions: Behavioral: HOP'N After-school Program

INTERVENTIONS:
Behavioral: HOP'N After-school Program — Daily 30 minutes of physical activity following CATCH guidelines, Daily healthful snack with fruit/vegetables, Weekly nutrition and physical activity education based on social cognitive theory.

SUMMARY:
This study presents evaluates the effectiveness of the Healthy Opportunities for Physical Activity(HOP'N) After-School Program on preventing obesity in children. The investigators hypothesized that normal and overweight/obese children attending after-school sites randomized to the control condition will increase in weight status to a greater extent compared to children at sites randomized to receive the HOP'N program. The investigators also hypothesized that after-school intervention HOP'N sites will increase in physical activity and healthful eating opportunities compared to control sites.

DETAILED DESCRIPTION:
The dramatic increase in the prevalence of overweight among children and adolescents has led to obesity prevention becoming a major national health priority. Although schools offer a logical choice for a setting to reach a great number of youth, these disappointing findings may be due in part to the difficulties of implementing interventions in school settings where competing demands for time have made it difficult to add anything other than academics to the school day. After-school programs may provide promise for preventing child obesity because there are fewer bureaucratic obstacles and curricular inflexibilities. A three-year group-randomized controlled trial will be conducted with random assignment at the school level . The study will use a nested cross section design with a baseline year, and two subsequent intervention years.

ELIGIBILITY:
Inclusion Criteria:

* after-school program participant in fourth grade group
* informed parental consent
* assent to participate in Body Mass Index assessment

Exclusion Criteria:

* third or fourth grade student
* participant in study in previous year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2005-08; Primary Completion 2008-05 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index Z-Score | Fall 2005, Spring 2006, Fall 2006, Spring 2007, Fall 2007, Spring 2008

SECONDARY OUTCOMES:
physical activity | Six times yearly

CONTACTS AND LOCATIONS:
Overall Officials: David A Dzewaltowski, Ph.D., Principal Investigator — Kansas State University
Locations (1):
- Kansas State University, Manhattan, Kansas, United States

REFERENCES:
- [Background] Geller KS, Dzewaltowski DA. Longitudinal and cross-sectional influences on youth fruit and vegetable consumption. Nutr Rev. 2009 Feb;67(2):65-76. doi: 10.1111/j.1753-4887.2008.00142.x. PMID 19178647
- [Result] Geller KS, Dzewaltowski DA. Examining elementary school--aged children's self-efficacy and proxy efficacy for fruit and vegetable consumption. Health Educ Behav. 2010 Aug;37(4):465-78. doi: 10.1177/1090198109347067. Epub 2009 Oct 26. PMID 19858314
- [Result] Geller KS, Dzewaltowski DA, Rosenkranz RR, Karteroliotis K. Measuring children's self-efficacy and proxy efficacy related to fruit and vegetable consumption. J Sch Health. 2009 Feb;79(2):51-7. doi: 10.1111/j.1746-1561.2008.00376.x. PMID 19187083
- [Result] Coleman KJ, Geller KS, Rosenkranz RR, Dzewaltowski DA. Physical activity and healthy eating in the after-school environment. J Sch Health. 2008 Dec;78(12):633-40. doi: 10.1111/j.1746-1561.2008.00359.x. PMID 19000239
- [Result] Trost SG, Rosenkranz RR, Dzewaltowski D. Physical activity levels among children attending after-school programs. Med Sci Sports Exerc. 2008 Apr;40(4):622-9. doi: 10.1249/MSS.0b013e318161eaa5. PMID 18317385
- [Derived] Virgara R, Phillips A, Lewis LK, Baldock K, Wolfenden L, Ferguson T, Richardson M, Okely A, Beets M, Maher C. Interventions in outside-school hours childcare settings for promoting physical activity amongst schoolchildren aged 4 to 12 years. Cochrane Database Syst Rev. 2021 Sep 27;9(9):CD013380. doi: 10.1002/14651858.CD013380.pub2. PMID 34694005
- [Derived] Rosenkranz RR, Welk GJ, Dzewaltowski DA. Environmental correlates of objectively measured physical activity and sedentary behavior in after-school recreation sessions. J Phys Act Health. 2011 Sep;8 Suppl 2:S214-21. PMID 21918235
- [Derived] Dzewaltowski DA, Rosenkranz RR, Geller KS, Coleman KJ, Welk GJ, Hastmann TJ, Milliken GA. HOP'N after-school project: an obesity prevention randomized controlled trial. Int J Behav Nutr Phys Act. 2010 Dec 13;7:90. doi: 10.1186/1479-5868-7-90. PMID 21144055